CLINICAL TRIAL: NCT01079559
Title: The Effectiveness of Antibiotic Cement Compared to Regular Cement in Reducing the Rate of Infection Following Total Knee Arthroplasty: The ABC Feasibility Study
Brief Title: The Effectiveness of Antibiotic Cement (ABC) Compared to Regular Cement in Reducing the Rate of Infection Following Total Knee Arthroplasty: The ABC Trial
Acronym: ABC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIHR-2010-222495
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Infection; Osteoarthritis of the Knee
Keywords: total knee arthroplasty; infection; antibiotic bone cement
MeSH Terms: conditions — Infections; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simplex™ P (Active Comparator): All patients will receive preoperative antibiotics administered within the hour prior to surgery. All patients will undergo a cemented total knee replacement (both femoral and tibial components) with the type of implant left to the discretion of the surgeon. The patella may or may not be resurfaced depending on indication and preference. All patients will receive one of the two study cements (Simplex™ P with Tobramycin or Simplex™ P) in a blinded fashion; all cement vials will be similar in size and shape and the cement will be similar in odour, color and texture. No additional antibiotics will be added to the cement. Surgeons can use their preferred cement preparation technique (i.e. manual or vacuum mixing). The use of a suction drain will depend on surgical indication and preference.
  Interventions: Device: Simplex™ P
- Simplex™ P with Tobramycin (Experimental): All patients will receive preoperative antibiotics administered within the hour prior to surgery.All patients will undergo a cemented total knee replacement (both femoral and tibial components) with the type of implant left to the discretion of the surgeon. The patella may or may not be resurfaced depending on indication and preference. All patients will receive one of the two study cements (Simplex™ P with Tobramycin or Simplex™ P) in a blinded fashion; all cement vials will be similar in size and shape and the cement will be similar in odour, color and texture. No additional antibiotics will be added to the cement. Surgeons can use their preferred cement preparation technique (i.e. manual or vacuum mixing). The use of a suction drain will depend on surgical indication and preference.
  Interventions: Device: Simplex™ P with Tobramycin

INTERVENTIONS:
Device: Simplex™ P with Tobramycin — All patients will receive preoperative antibiotics administered within the hour prior to surgery.All patients will undergo a cemented total knee replacement (both femoral and tibial components) with the type of implant left to the discretion of the surgeon. The patella may or may not be resurfaced depending on indication and preference. All patients will receive one of the two study cements (Simplex™ P with Tobramycin or Simplex™ P) in a blinded fashion; all cement vials will be similar in size and shape and the cement will be similar in odour, color and texture. No additional antibiotics will be added to the cement. Surgeons can use their preferred cement preparation technique (i.e. manual or vacuum mixing). The use of a suction drain will depend on surgical indication and preference.
  Arms: Simplex™ P with Tobramycin
Device: Simplex™ P — All patients will receive preoperative antibiotics administered within the hour prior to surgery.All patients will undergo a cemented total knee replacement (both femoral and tibial components) with the type of implant left to the discretion of the surgeon. The patella may or may not be resurfaced depending on indication and preference. All patients will receive one of the two study cements (Simplex™ P with Tobramycin or Simplex™ P) in a blinded fashion; all cement vials will be similar in size and shape and the cement will be similar in odour, color and texture. No additional antibiotics will be added to the cement. Surgeons can use their preferred cement preparation technique (i.e. manual or vacuum mixing). The use of a suction drain will depend on surgical indication and preference.
  Arms: Simplex™ P

SUMMARY:
Rationale: Infection following total knee replacement (TKA) is a devastating complication that usually requires prosthesis removal, hospitalization while the infection is eradicated, and a second surgery to implant a revision prosthesis. For primary TKA, prophylactic antibiotic-loaded cement (ABC) may not only reduce the rate of infection it may also reduce the rate of revisions due to implant loosening. Current controversy about the use of ABC exists around the world. Without a definitive trial, patients will be exposed to a treatment of uncertain efficacy that may cause antibiotic resistant bacterial strains and will certainly generate high costs to the healthcare system. Purpose: To determine, 1) the extent to which ABC compared to regular cement reduces the infection rate in patients over the first two years following TKA and, 2) the resource use implications associated with the use of ABC for TKA. Methods: This is a randomized clinical trial in which 8,800 patients with undergoing primary TKA are allocated to either Simplex™ P with Tobramycin or Simplex™ P bone cement. We will exclude patients with a prior joint infection, an allergy to tobramycin, and those with no fixed address. All patients will be administered IV antibiotics immediately prior to surgery. Patients and surgeons will be blind to group allocation. The primary outcome measure is infection. Follow-up visits will take place at 6 weeks and 3, 12 and 24 months postoperative. A blinded adjudicator will review all reported infections and determine whether the putative infection is a study event. Blinded radiologists will interpret the 2 year series of radiographs for each patient. We will compare the rates of infection and implant loosening between the two treatment groups using survival analyses. This study includes a full economic analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with osteoarthritis of the knee,
* patients who are undergoing primary knee replacement,
* patients who are able to provide informed consent.

Exclusion Criteria:

* patients with a prior joint infection,
* patients who have a known allergy to tobramycin, and
* patients who have no fixed address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
relative risk of infection | 6 weeks and 3, 12 and 24 months postoperative
  patients suspected of having an infected total knee replacement in the post-operative period will be evaluated clinically, and will undergo lab evaluation and an aspiration

SECONDARY OUTCOMES:
radiographic evidence of prosthetic failure | 6 weeks and 3, 12 and 24 months postoperative
patient-reported disease-specific health-related quality of life (HRQOL) | 6 weeks and 3, 12 and 24 months postoperative
cost-effectiveness | 6 weeks and 3, 12 and 24 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Bryant, PhD, Principal Investigator — Western University, Canada; Steven J MacDonald, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada